CLINICAL TRIAL: NCT01078727
Title: Thermal Stimulation on Upper Extremity Movement and Function in Patients With Stroke
Brief Title: Safety Study of Thermal Stimulation on Upper Extremity Motor Recovery to Stroke
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other); National Taiwan University (Other); Kaohsiung Medical University (Other)
Responsible Party: Jau-Hong Lin/Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUH-IRB-950320
Record Dates: First submitted 2010-02-11; First posted 2010-03-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2008-02

CONDITIONS: Stroke
Keywords: Thermal Stimulation; Upper Extremity; Motor Recovery; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: A custom-made constant temperature thermal stimulation system (FIRSTEK, Model-B401L, B-300, local company, Taiwan). — The subjects meeting our criteria will be randomly assigned to either the experimental group or the control group. First stage (3 months after onset), the subjects in the experimental group will receive an upper extremity Thermal Stimulation (TS) protocol for 30 minutes (3 times a week for 8 weeks). The subjects in the control group will receive a lower extremity TS protocol.

SUMMARY:
Improving upper extremity movement and function in patients with stroke has been one of the primary goals for patients and rehabilitation professionals. Thermal stimulation (TS) had been first found by a domestic research group to be effective to facilitate sensory and motor recovery in patients with stroke within a month. However, the immediate and long-term effects of TS and the mechanism of brain plasticity in patients with stroke for more than three months (golden recovery stage) remain unknown. Thus, we will design a single-blind randomized controlled trial to investigate the immediate and long-term effects of TS in patients with stroke at subacute and chronic stages.

DETAILED DESCRIPTION:
The study was an assessor-blinded randomized controlled clinical trial. Participants with UE impairment for more than 3 months poststroke were randomly assigned to either the experimental (EXP) group or the control group. All participants received regular conventional rehabilitation programs. The EXP group received an additional UE-TS protocol for 30 minutes a day (3 days/week for 8 weeks); the control group received the same TS protocol over the lower extremity (LE). The Brunnstrom's recovery stage, the Modified Ashworth Scale (MAS), the Stroke Rehabilitation Assessment of Movement (STREAM), the Action Research Arm Test (ARAT), and the Barthel Index (BI) were outcome measures and were administered at baseline, 4 weeks and 8 weeks post inception, and at one-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. first-ever stroke survivors with unilateral hemispheric lesions from a hemorrhagic or nonhemorrhagic stroke;
2. stroke onset more than 3 months and less than 3 years prior to study enrollment;
3. no severe cognitive impairments and able to follow instructions;
4. the ability to sit on a chair for more than 30 minutes independently.

Exclusion Criteria:

1. musculoskeletal or cardiac disorders that could potentially interfere with experimental tests;
2. diabetic history or sensory impairment attributable to peripheral vascular disease or neuropathy;
3. speech disorder or global aphasia;
4. participating in any experimental rehabilitation or drug studies;
5. skin injuries, burns, or fresh scars at the sites of stimulation;
6. contraindication of heat or ice application.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Stroke Rehabilitation Assessment of Movement | 3 months
Action Research Arm Test | 3 months
Barthel Index | 3 months
Modified Ashworth Scale | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: J H Lin, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Department of Physical Therapy, Kaohsiung Medical University, Kaohsiung City, Taiwan